CLINICAL TRIAL: NCT06469216
Title: Efficacy of Hyaluronic Acid in Prevention of Acute Radiation Proctitis: Multi-center, Double-blind, Randomized Controlled Trial
Brief Title: Efficacy of Hyaluronic Acid in Prevention of Acute Radiation Proctitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Gamal El Sheikh, Clinical pharmacist at Al-Ahrar Oncology Center, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-2023-018
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Radiation Proctitis; Acute Radiation Enteritis
Keywords: double blind; placebo control; Randomized Clinical Trial
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30 ml of Hyaluronic Acid (HA) enema will be given to the patients (Active Comparator): All patients will be prospectively randomized into two groups; either the treatment (HA) group or the control group. In this study protocol, 30 ml of HA enema and 30 ml of placebo enema (identical to treatment group enema but without HA) will be given to the patients as they lie on their left side with their right knee pulled up to the chest.
  Interventions: Drug: Hyaluronic Acid
- 30 ml of placebo enema (identical to treatment group enema but without HA) will be given to patients (Placebo Comparator): All patients will be prospectively randomized into two groups; either the treatment (HA) group or the control group. In this study protocol, 30 ml of HA enema and 30 ml of placebo enema (identical to treatment group enema but without HA) will be given to the patients as they lie on their left side with their right knee pulled up to the chest.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hyaluronic Acid — Hyaluronic Acid to be used as sodium hyaluronate powder plus inactive ingredient (Carboxy methyl cellulose) and to be dissolved in distilled water
  Other Names: Sodium Hyaluronate
  Arms: 30 ml of Hyaluronic Acid (HA) enema will be given to the patients
Other: Placebo — Inactive ingredient (Carboxy methyl cellulose) to be used as powder and to be dissolved in distilled water
  Arms: 30 ml of placebo enema (identical to treatment group enema but without HA) will be given to patients

SUMMARY:
A randomized placebo-controlled clinical trial to evaluate efficacy of hyaluronic acid in prevention of acute radiation proctitis among oncology patient population especially who are diagnosed with abdomeno-pelvic tumors and subsequently required radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with pelvic or gastrointestinal malignancies (tumors in uterus, cervix, prostate, seminal vesicles, kidney, colon, etc.),
* All patients who required adjuvant or radical radiation therapy;
* Age < 80 years;
* Karnofsky Performance Status ≥ 60

Exclusion Criteria:

* Patients were excluded if they had

  * gt; previous pelvic radiotherapy,
  * gt; inflammatory bowel disease or
  * gt; rectal issues (e.g., haemorrhoids).
* Patients diagnosed with cancer rectum

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Time (in days) to occurrence of Acute Radiation Proctitis | for each patient: time from the first day of radiation therapy for up to 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Maher teaching hospitals, Cairo, Cairo Governorate
  - Al-Ahrar teaching hospital, Zagazig, Sharqia Province